CLINICAL TRIAL: NCT05548998
Title: Effect of Low Fresh Gas Flow Volatile Anesthetics on Postoperative Neurocognitive Function in Elderly Patients
Brief Title: Effect of Low Flow Anesthetics on Neurocognitive Decline in the Elderly
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Namigar Turgut, Professor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 1206
Record Dates: First submitted 2022-09-17; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Neurocognitive Disorders; Inhalation; Vapor
MeSH Terms: conditions — Neurocognitive Disorders; Respiratory Aspiration | interventions — Anesthesia, General; Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High flow cohort (HFA): Patients, whose maintenance phase of anesthesia is managed with a fresh gas flow ≥ 1L/min, were included in this cohort.
  Interventions: Other: General anesthesia with high fresh gas flow; Diagnostic Test: Mini mental state examination; Diagnostic Test: Visual Analogue Scale
- Low flow cohort (LFA): Patients, whose maintenance phase of anesthesia is managed with a fresh gas flow < 1L/min, were included in this cohort.
  Interventions: Other: General anesthesia with low fresh gas flow; Diagnostic Test: Mini mental state examination; Diagnostic Test: Visual Analogue Scale

INTERVENTIONS:
Other: General anesthesia with low fresh gas flow — General anesthesia with a fresh gas flow lower than 1L/min for the maintenance phase of anesthesia
  Groups: Low flow cohort (LFA)
Other: General anesthesia with high fresh gas flow — General anesthesia with a fresh gas flow equal to or higher than 1L/min for the maintenance phase of anesthesia
  Groups: High flow cohort (HFA)
Diagnostic Test: Mini mental state examination — 6 category and 30-point test to inquire patient's cognitive function
  Other Names: MMSE
Diagnostic Test: Visual Analogue Scale — The patient's self-reported pain intensity according to a visual scale between 0 and 100
  Other Names: VAS

SUMMARY:
This study aims to investigate the effect of inhaled anesthetics with a low fresh gas flow on cognitive function of elderly patients undergoing elective surgery

DETAILED DESCRIPTION:
Geriatric patients scheduled to undergo surgery were tested with Mini Mental State Examination (MMSE) in the preoperative visit. MMSE was repeated postoperatively at the 6th hour, the 1st, 3rd, and 7th day. Visual analogue scale (VAS) test was performed simultaneously on the postoperative 6th hour, the 1st, 3rd, and 7th day. Two cohorts were created according to the amount of fresh gas flow (low flow vs high flow) in the maintenance phase of the inhalational anesthetic. MMSE scores were compared between cohorts and baseline. VAS scores were compared between cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Age>65
* Consenting to participate
* Scheduled for surgery longer than 2 hours under GA
* Able to read and write

Exclusion Criteria:

* Age<65
* Refusing to participate
* Existing visual impairment preventing the patient from reading or writing
* Unable to read and write
* Existing major neurocognitive disorder
* Use of TIVA or regional techniques
* Allergies to the volatile agents
* Uncontrolled DM, acute alcohol intoxication
* Conditions increasing tissue oxygen consumption (sepsis, thyrotoxicosis, etc.)
* Anticipation/existence of major hemorrhage
* Haemodynamic instability > 10 min or more than 5 times intraoperatively

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Cohorts were selected from geriatric patients (>65 y.o.) of a tertiary care clinic who underwent surgery under general anesthesia with different fresh gas flows for the maintenance phase.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in neurocognitive status on the 30 point MMSE at postoperative 24th hour | Baseline and postoperative day 1
  A Mini-Mental State Examination (MMSE) is a set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory).

SECONDARY OUTCOMES:
Change from baseline in neurocognitive status on the 30 point MMSE at postoperative 6th hour | Baseline and postoperative hour 6
  A Mini-Mental State Examination (MMSE) is a set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory).
Change from baseline in neurocognitive status on the 30 point MMSE at postoperative 3rd day | Baseline and postoperative day 3
  A Mini-Mental State Examination (MMSE) is a set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory).
Change from baseline in neurocognitive status on the 30 point MMSE at postoperative 7th day | Baseline and postoperative day 7
  A Mini-Mental State Examination (MMSE) is a set of 11 questions that doctors and other healthcare professionals commonly use to check for cognitive impairment (problems with thinking, communication, understanding and memory).
Change from baseline in pain on the 10 point VAS scale at postoperative 6th hour | Baseline and postoperative hour 6
  The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge
Change from baseline in pain on the 10 point VAS scale at postoperative 24th hour | Baseline and postoperative hour 24
  The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge
Change from baseline in pain on the 10 point VAS scale at postoperative 3rd day | Baseline and postoperative day 3
  The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge
Change from baseline in pain on the 10 point VAS scale at postoperative 7th day | Baseline and postoperative day 7
  The visual analog scale (VAS) is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge

CONTACTS AND LOCATIONS:
Overall Officials: Namigar TURGUT, Principal Investigator — Prof. Dr. Cemil Taşcıoğlu City Hospital
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No